CLINICAL TRIAL: NCT02158416
Title: Blinded Study on Consecutive Transfusable Platelet Products Tested With the ThromboLUX® Platelet Quality Test
Brief Title: Platelet Products Tested With the ThromboLUX® Platelet Quality Test
Status: Completed | Type: Observational
Sponsor: LightIntegra Technology (Industry)
Responsible Party: Sponsor
Other Study IDs: TLXPRO017
Record Dates: First submitted 2014-03-17; First posted 2014-06-06 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Poor Platelet Transfusion Outcome
Keywords: platelet; transfusion; ThromboLUX; corrected count increment; thrombocytopenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hematology-oncology: hematology-oncology outpatients requiring platelet transfusion

SUMMARY:
The planned minimal risk study is a blinded study on consecutive transfusable platelet products. The aim of the study is to evaluate the quality of platelet components sampled prior to transfusion.

The primary patient transfusion outcome in this study is the 1-hour corrected count increment (1 hr CCI), which is a widely accepted clinical outcome measure. Platelet products will be sampled for ThromboLUX testing before being sent from the blood bank to the treatment center. After receipt at the treatment center, the platelet products will be used as per regular clinical practice, and the outcome data from each patient will be collected. At the end of the study, TLX Scores will be compared to the transfusion outcomes to determine if a low TLX Score is associated with a poor transfusion outcome.

During the course of the study, the TLX Score will not be known to the clinicians, or utilized in any way to decide if the platelet product should be transfused.

ELIGIBILITY:
Inclusion Criteria:

* adult hematology-oncology outpatients
* stable and thrombocytopenic

Exclusion Criteria:

* age <18 yrs
* splenomegaly
* unable to provide informed consent
* pregnancy
* acute promyelocytic leukemia
* ITP (Idiopathic thrombocytopenic purpura)
* HUS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adults who require treatment of a blood cancer with platelet transfusion(s). Patients will be stable and thrombocytopenic, however treatment center will intervene for bleeding. Adult hematology-oncology outpatients.
Sampling Method: Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2013-12; Primary Completion 2014-07 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
TLX Score Correlation with CCI | Patients are expected to be enrolled for an average of 6 months.
  The value of the ThromboLUX Score (obtained from platelet products with the ThromboLUX platelet quality test system) to predict patient transfusion outcome (measured as 1hr corrected count increment CCI). The correlation between ThromboLUX score and 1hr CCI (study endpoint) will be reported at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: William A Heaton, MD, Principal Investigator — Northwell Health
Locations (1):
- Monter Center, New Hyde Park, New York, United States